CLINICAL TRIAL: NCT04344236
Title: A Phase II, Randomized, Open-label, Single-institution Study of the Effects of Povidone Iodine Oral Gargles and Nasal Rinses on Viral Load in Patients With COVID-19
Brief Title: Gargling and Nasal Rinses to Reduce Oro- and Nasopharyngeal Viral Load in Patients With COVID-19
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was withdrawn by the institution to minimize risk to patients and staff with regard to COVID-19.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: s20-00444
Record Dates: First submitted 2020-04-08; First posted 2020-04-14 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Povidone

STUDY DESIGN:
Intervention Model Description: Randomized controlled open label trial, parallel design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Control (No Intervention)
- Saline oral/nasal rinse (Experimental)
  Interventions: Drug: Saline oral/nasal rinse
- 0.5% Povidone/Iodine oral/nasal rinse (Experimental)
  Interventions: Drug: 0.5% Povidone/Iodine oral/nasal rinse
- 0.12% Chlorhexidine oral/nasal rinse (Experimental)
  Interventions: Drug: 0.12% Chlorhexidine oral/nasal rinse

INTERVENTIONS:
Drug: Saline oral/nasal rinse — 5 cc of nasal rinses total for both nostrils + 20 cc of oral gargles, 4 times a day, for 7 days.
  Arms: Saline oral/nasal rinse
Drug: 0.5% Povidone/Iodine oral/nasal rinse — 5 cc of nasal rinses total for both nostrils + 20 cc of oral gargles, 4 times a day, for 7 days.
  Arms: 0.5% Povidone/Iodine oral/nasal rinse
Drug: 0.12% Chlorhexidine oral/nasal rinse — 5 cc of nasal rinses total for both nostrils + 20 cc of oral gargles, 4 times a day, for 7 days.
  Arms: 0.12% Chlorhexidine oral/nasal rinse

SUMMARY:
For this study, 48 patients who have been diagnosed with COVID-19 will be randomly assigned to four study groups: control, saline, chlorhexidine gluconate, and povidone-iodine. Each patient will be asked to gargle with a solution of either saline, chlorhexidine gluconate, or povidone-iodine or nothing (control group) as well as spray the same solution in their nose four times daily. Patients will then be tested for COVID-19 once daily in the evening for 7 days and viral loads will be measured.

DETAILED DESCRIPTION:
COVID-19 has emerged as a worldwide pandemic and there is a strong need for identification of any measures that can be used to treat this illness or reduce its transmission from person to person. Povidone-iodine has been shown to have virucidal properties against multiple viruses including against the virus that causes SARS which is very similar in makeup to the virus causing COVID-19.

The investigators hypothesize that 4x daily use of oral gargles and nasal rinses using a povidone iodine solution will help to reduce the viral load in the nasopharynx and oropharynx in patients who are COVID-19+. If this hypothesis is shown to be true this could potentially have an impact on time to recovery of clinical symptoms as well as reduce shedding of the virus by infected patients. A time course of 7 days was chosen in order to recognize a trend in the viral load over time for patients receiving each of the interventions. Chlorhexidine gluconate and saline rinses were chosen as additional treatment arms as these are frequently used for oral and nasal hygiene and their role in affecting viral load is currently unknown.

ELIGIBILITY:
Inclusion Criteria:

1. Positive test for COVID-19
2. Age 18-79 years
3. Willing and able to perform oral gargles and nasal rinses four times daily

Exclusion Criteria

1. Requiring mechanical ventilation
2. Unable or unwilling to perform oral gargles and nasal rinses four times daily
3. History of chronic upper respiratory tract disease
4. Known iodine allergy
5. History of thyroid disease

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04-09 (Actual); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-05-09 (Estimated)

PRIMARY OUTCOMES:
Viral load (and/or cycle time to PCR as a proxy for quantitative viral load) in the nasopharynx and oropharynx | 7 days
  nasopharyngeal swab for viral PCR will be taken at the end of each day for 7 days

SECONDARY OUTCOMES:
Oxygen requirement of the patient | 7 days
  Recorded daily
Oxygen saturation of the patient | 7 days
  Recorded daily

CONTACTS AND LOCATIONS:
Overall Officials: Scott Rickert, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: [contact information for PI or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: Requests should be directed to scott.rickert@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.